CLINICAL TRIAL: NCT01690078
Title: Predictive Modeling for Treatment of Upper Airway Obstruction in Young Children
Brief Title: Functional Modeling of the Pediatric Airway
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-1634; R01HL105241 (NIH)
Record Dates: First submitted 2012-07-30; First posted 2012-09-21 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2016-06

CONDITIONS: Subglottic Stenosis (SGS); Pierre Robin Sequence (PRS); Micrognathia; Normal Controls From CT Scans of the Upper Airway
Keywords: Airway modeling; Pierre Robin Sequence or PRS; Micrognathia; Subglottic Stenosis or SGS
MeSH Terms: conditions — Pierre Robin Syndrome; Micrognathism; Prieto X-linked mental retardation syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cross sectional: Cross sectional study where subjects with PRS, micrognathia, or SGS will have a single study visit that will be scheduled within 14 days of a clinically indicated upper airway endoscopy. CT scans of the neck or maxillofacial CT will be obtained in all subjects. During upper airway endoscopy, airway measurements will be conducted. Cohort may include subjects who have previously undergone medical or surgical intervention for their airway obstruction, or who are currently undergoing multidisciplinary team management. The following data will be collected: clinical parameters, Obstructive Sleep Apnea (OSA)OSA-18 (quality of life) questionnaire, and lung function tests (subjects > 4 years of age). Clinically indicated swallowing studies and voice evaluations will be collected.
- Longitudinal: The prospective, longitudinal cohort arm of the study is designed to describe the effects of treatment on clinical and computational model endpoints. This is performed in a subset of subjects with PRS, micrognathia, or SGS who are scheduled for clinically indicated upper airway endoscopy and who are scheduled to complete a definitive treatment course which necessitates multiple endoscopic evaluations and follow-up imaging. Subjects will have an entry visit comparable to the cross-sectional entry visit. Longitudinal subjects will have up to 3 additional study visits over a 12 to 15-month period.
- Normal Control Data: Normal de-identified control data is retrospectively collected from clinically indicated CT scans of the neck and maxillofacial CT scans in children less than 18 years of age.

SUMMARY:
The investigators hypothesize that a functional computational model that simulates the mechanical and aerodynamic behavior of the upper airway in children with Pierre Robin Sequence (PRS) and laryngeal lesions (e.g. subglottic stenosis or SGS) can be used as an effective diagnostic and treatment planning tool.

ELIGIBILITY:
Inclusion Criteria:

1. Micrognathia, Suspected or Diagnosis of PRS, defined (Gorlin) as:

   micrognathia (mandibular hypoplasia), cleft palate and airway obstruction, and/or

   Diagnosis of SGS defined (Bluestone) as:
   * subglottic airway diameter of 4 mm or less in a term neonate;
   * subglottic airway diameter of 3.5 mm or less in a premature neonate;
   * inability to pass an endotracheal tube of expected size for age
2. Informed consent by parent or legal guardian
3. Age < 18 years at enrollment
4. Scheduled for clinically indicated endoscopic upper airway evaluation
5. Ability to comply with study visits and study procedures as judged by the site investigator

Inclusion criterion also included for Specific Aim 2 (Longitudinal):

Subjects must be scheduled for an operative procedure to correct or bypass upper airway obstruction (i.e. mandibular distraction, endoscopic airway surgery, laryngotracheoplasty, cricotracheal resection, or tracheostomy) OR recently (within past 4 weeks) diagnosed as having an anomaly not currently requiring surgical management.

Exclusion Criteria:

1. Acute, intercurrent respiratory infection, defined as an increase from baseline in cough, wheezing, or respiratory rate with onset in the preceding week.
2. Physical findings at screening that would compromise the safety of the participant or the quality of the study (i.e. fever, increased respiratory rate above baseline, significant acute emesis, or alteration in baseline neurologic status).
3. For research CT scans any sedation risk, such as Bronchopulmonary Dysplasia (BPD) with upper airway obstruction, residual oxygen requirement, and an unsecured airway.

Control data will be collected from clinically indicated neck or maxillofacial CT imaging data that include the entire airway with no noted airway obstructions or airway abnormalities.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children < 18 years of age with a diagnosis of either Pierre Robin Sequence, Micrognathia or Subglottic Stenosis.
  Clinically indicated control data will be collected from CT scans of neck and maxillofacial CT scans performed on children < 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Functional computational model outcome parameters | years 1- 3
  Change in functional computational modeling parameters as compared to the change in percent of total time spent with oxygen saturation < 90% as noted on polysomnogram (physiologic measure) and change in airway measurements obtained via clinically indicated upper airway endoscopy (anatomic measure) pre and post-intervention(medical or surgical)

SECONDARY OUTCOMES:
Validation of Computational model | year 4
  Apply the computational model to infants and children being evaluated for Pierre Robin Sequence and Subglottic Stenosis, to determine the ability of the model to accurately predict the results of various potential interventions on anatomic and physiologic metrics.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie D Davis, MD, Principal Investigator — Indiana University School of Medicine; Carlton Zdanski, MD, Principal Investigator — University of North Carolina, Chapel Hill; Richard Superfine, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- North Carolina Children's Hospital, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Calloway HE, Kimbell JS, Davis SD, Retsch-Bogart GZ, Pitkin EA, Abode K, Superfine R, Zdanski CJ. Comparison of endoscopic versus 3D CT derived airway measurements. Laryngoscope. 2013 Sep;123(9):2136-41. doi: 10.1002/lary.23836. PMID 24167819
- [Background] Mitran S. Continuum-kinetic-microscopic model of lung clearance due to core-annular fluid entrainment. J Comput Phys. 2013 Jul 1;244:193-211. doi: 10.1016/j.jcp.2013.01.037. PMID 23729842
- [Background] Mitran (2012c), Predictive Modeling of Upper Airway Flow in Young Children, Proceedings, 34th Annual International Conference of the IEEE Engineering in Medicine and Biology Society (EMBC'12), San Diego, CA, (accepted).
- [Background] Mitran, S. (2012b), "Lattice Fokker-Planck Method Based on Wasserstein Gradient Flows", Phys. Rev.E., (under review).
- [Background] Alabi OS, Wu X, Harter JM, Phadke M, Pinto L, Petersen H, Bass S, Keifer M, Zhong S, Healey C, Taylor RM 2nd. Comparative Visualization of Ensembles Using Ensemble Surface Slicing. Proc SPIE Int Soc Opt Eng. 2012 Jan 22;8294:82940U. doi: 10.1117/12.908288. PMID 23560167
- [Background] Yi Hong, Yundi Shi, Martin Styner, Mar Sanchez, and Marc Niethammer. Simple Geodesic Regression for Image Time-Series. Accepted to the 5th Workshop on Biomedical Image Registration. 2012.
- [Background] Hong Y, Joshi S, Sanchez M, Styner M, Niethammer M. Metamorphic geodesic regression. Med Image Comput Comput Assist Interv. 2012;15(Pt 3):197-205. doi: 10.1007/978-3-642-33454-2_25. PMID 23286131
- [Background] Zdanski, C., Kimbell, J.S., Superfine, R.S., and Davis, S. (2012). Computational Fluid Dynamics Modeling of the Pediatric Airway Utilizing Computed Tomography in Children with Pierre Robin Sequence. Poster presentation, European Society of Pediatric Otolaryngology, Amsterdam, The Netherlands, May 20-23, 2012.